CLINICAL TRIAL: NCT06562985
Title: A Single Dose Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BAY 3018250 After Intravenous Infusion in Healthy Male Japanese Participants in a Dose Escalation Design and a Single Intravenous Bolus Injection in Healthy Adult Participants
Brief Title: A Study to Learn About How Safe BAY3018250 is and What Happens to it in Healthy Japanese Men and Adult Participants Aged 18 to 55 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22497
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Venous and Arterial Thrombotic and Thromboembolic Events; Healthy Volunteers
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose step 1 (Part A) (Experimental): Participants will receive a single dose of BAY3018250 dose step 1 via infusion in part A.
  Interventions: Drug: BAY3018250 Dose 1
- Dose step 2 (Part A) (Experimental): Participants will receive a single dose of BAY3018250 dose step 2 via infusion in part A.
  Interventions: Drug: BAY3018250 Dose 2 infusion
- Placebo (Part A) (Placebo Comparator): Participants will receive a single dose of BAY3018250 matching placebo via infusion in part A.
  Interventions: Drug: Placebo
- Dose step 2 (Part B) (Experimental): Participants will receive a single dose of BAY3018250 dose step 2 via injection in part B.
  Interventions: Drug: BAY3018250 Dose 2 injection
- Placebo (Part B) (Placebo Comparator): Participants will receive a single dose of BAY3018250 matching placebo via injection in part B.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY3018250 Dose 1 — Infusion, single dose
  Arms: Dose step 1 (Part A)
Drug: Placebo — BAY3018250 matching placebo, infusion
  Arms: Placebo (Part A)
Drug: Placebo — BAY3018250 matching placebo, injection
  Arms: Placebo (Part B)
Drug: BAY3018250 Dose 2 infusion — Infusion, single dose
  Arms: Dose step 2 (Part A)
Drug: BAY3018250 Dose 2 injection — Injection, single dose
  Arms: Dose step 2 (Part B)

SUMMARY:
Researchers are looking for a better way to treat people who have acute venous and arterial thrombotic and thromboembolic events. These are severe medical problems due to blood clots forming in and blocking blood vessels.

The study treatment BAY3018250 is under development to treat acute venous and arterial thrombotic and thromboembolic events. It aims to work by dissolving blood clots in the blood vessels.

In this study, participants will be healthy and will not benefit from receiving BAY3018250. However, the study will provide information on how to test BAY3018250 in future studies in people with acute venous and arterial thrombotic and thromboembolic events.

During the study, researchers will use two different methods of giving BAY3018250 to participants. This may help in developing a faster method of giving this treatment in case of emergencies.

The main purpose of this study is to check how safe BAY3018250 is and if it is well tolerated by participants. For this, researchers will study the number and severity of medical problems in:

* healthy Japanese men after receiving different doses of BAY3018250 as an infusion into a vein.
* healthy adult participants after receiving a certain dose of BAY3018250 by an injection.

These medical problems are also known as "adverse events". Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatment.

This study will have two parts: Part A and Part B:

- Only healthy Japanese men can join Part A of the study, which will have two groups. In the first group, participants will receive a low dose of BAY3018250. If researchers consider this dose to be safe, the next group will receive a higher dose.

In each group, participants will be randomly assigned to receive BAY3018250 or placebo as an infusion into a vein once during the study. A placebo looks like a study drug but does not have any medicine in it.

- Healthy men and women can join Part B of the study. Participants will be randomly assigned to receive a certain dose of BAY3018250 or placebo by an injection once during the study.

Each participant will be in the study for around 14 weeks, which includes:

* a visit to the hospital within 3 weeks of taking any treatment to confirm if the participant can take part in the study
* a hospital stay of 1 week, during which participants will receive their assigned treatment, have blood and urine tests and complete health check-ups
* six follow-up visits to the hospital until about 11 weeks after receiving the study treatments During the study, the doctors and their study team will check participants' health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram (ECG) As this study is conducted in healthy participants who will not benefit from the treatment, access to the treatment after the study is not planned.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

Part A:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, safety laboratory tests, vital signs, and electrocardiogram (ECG).
* Japanese who was born in Japan and whose parents and grandparents must have been Japanese and who has not lived outside of Japan for more than 10 years and has not significantly modified their diets since leaving Japan.
* Male

Part B:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, safety laboratory tests, vital signs, and ECG.
* Male or female (postmenopausal or hysterectomized only)

Exclusion Criteria:

* Medical disorder, condition (e.g., after surgical procedure), or history of such that would impair the participant's ability to take part in or complete this study in the opinion of the investigator. This includes family history indicating hereditary predisposition of relevant diseases and history of non- persisting diseases with possible impact on study participation.
* Increased bleeding risk: known coagulation disorders (e.g., von Willebrand´s disease, hemophilia), periodontitis, symptomatic hemorrhoids, acute gastritis, peptic ulcer, or similar diseases with tendency to lead to bleedings, known sensitivity to common causes of bleeding (e.g., nasal, etc.), or history of hemorrhage and gastrointestinal ulceration within 6 months prior to the screening visit.
* Family history of hereditary or not explainable bleeding disorders.
* History of thrombosis or family history of hereditary or not explainable diseases with increased risk for thrombosis or thromboembolic events.
* Tendency of easy bruising.
* Platelets out of reference range.
* Activated partial thromboplastin time (aPTT) or prothrombin time (PT) out of reference range.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced treatment-emergent adverse events (TEAEs) after administration of BAY3018250 | Administration of study intervention until last follow-up visit (75 days)

SECONDARY OUTCOMES:
Cmax of BAY3018250 | Administration of study intervention until Day 75
AUC of BAY3018250 | Administration of study intervention until Day 75
  If AUC cannot be determined reliably in all participants, AUC(0-tlast) will be used instead.

CONTACTS AND LOCATIONS:
Locations (1):
- Collaborative Neuroscience Research, LLC, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22497